CLINICAL TRIAL: NCT02110537
Title: Clinical Trial to Evaluate the Antiarrhythmic Effects of Acupuncture for Drug Resistant Persistent Atrial Fibrillation: Randomized, Participant and Assessor Blinded, Sham-controlled, Clinical Trial
Brief Title: Acupuncture in Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Weon Kim, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HI13C0580
Record Dates: First submitted 2014-04-06; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Acupuncture; Recurrence; Electrical cardioversion
MeSH Terms: conditions — Atrial Fibrillation; Recurrence | interventions — Flecainide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Acupuncture + flecainide (Experimental): The participants in this group receive verum acupuncture treatment once a week for 10 weeks and flecainide 75 mg twice daily.
  Interventions: Procedure: Active Acupuncture; Drug: flecainide
- Sham acupuncture + flecainide (Sham Comparator): The participants in this group receive sham acupuncture treatment once a week for 10 weeks and flecainide 75 mg twice daily.
  Interventions: Procedure: Sham acupuncture; Drug: flecainide

INTERVENTIONS:
Procedure: Active Acupuncture — Active acupuncture treatment group consists of electroacupuncture (EA) and intradermal acupuncture (IDA). For EA treatment, unilateral PC5, PC6, ST36, and ST37 are chosen. Disposable, sterile needles and low frequency electrical stimulator (ES-160, ITO, Japan) are used. Each needle is inserted to the depth of 2 ± 0.5 cm with a 90 degree angle. Thereafter, needles are connected with the pole and electrical stimulation is applied with 2Hz, continuous wave current for 20 minutes. For IDA treatment, bilateral HT7 and TF4 are selected. Disposable, sterile, sticker-type needles (0.18 mm x 1.3 mm x 1.5mm) are used. Attached needles are maintained as long as possible.
  Arms: Active Acupuncture + flecainide
Procedure: Sham acupuncture — For sham intervention, nonacupuncture points are used. As with active treatment group, two types of acupuncture, sham EA and sham IDA, compose the sham intervention. Electrical acupuncture is connected but electrical stimulation is not given to sham acupuncture group.
  Arms: Sham acupuncture + flecainide
Drug: flecainide — Both groups commonly take antiarrhythmic medication (flecainide 75 mg twice daily) during study period. Flecainide administration is initiated 2 weeks before electrical cardioversion and maintain during follow up period.
  Other Names: tambocor

SUMMARY:
The aim of this trial is to evaluate the effect of acupuncture on prevention of atrial fibrillation (AF) recurrence after electrical cardioversion (EC) for persistent AF patients resistant to the antiarrhythmic drugs (AADs).

DETAILED DESCRIPTION:
This is a multicenter, prospective, participant and assessor blinded, randomized, sham-controlled clinical trial with 2 parallel arms. To evaluate the efficacy and safety of acupuncture, a total of 80 persistent AF participants will be recruited and randomly assigned to active acupuncture and sham acupuncture group. Both group commonly take antiarrhythmic medication during study period. These patients who are resistant to drug therapy will get a electrical cardioversion. After cardioversion, the recurrence rate and duration of atrial fibrillation free time will be evaluated.

This trial consists of 2 weeks of observation and medical therapy, 2 weeks of acupuncture intervention before EC, EC and acupuncture intervention, 7 weeks of additional intervention, and 5 weeks of follow-up. After randomization, participants receive 10 sessions of acupuncture treatments over 10 weeks. The outcome is assessed at 2, 4, 6, 8, and 16 week after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Persistent AF lasting ≥ 7 days
* Ages in 20-75 years
* Resistant with antiarrhythmic drugs
* Written informed consent

Exclusion Criteria:

* Age below 20 years or above 75 years
* Severe valvular heart disease
* History of open heart surgery
* History of treatment for myocardial infarction (MI) within recent 6 weeks
* Patients under or requiring the administration of antiviral drugs
* 2nd degree atrioventricular block or more than two fascicular block
* Severe pulmonary, liver, or renal disease
* Previous acupuncture treatment for cardiovascular condition within 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation evaluated on serial electrocardiography and 48 hour holter monitoring after sinus conversion by electrical cardioversion | 3 months after electrical cardioversion
  When patient feel symptoms such as palpitation and chest discomfort, the patients are recommended to visit hospital to check out the recurrence of atrial fibrillation.

SECONDARY OUTCOMES:
Changes in function and volume of left atrium and left atrial appendage evaluated by echocardiography | 3 months after electrical cardioversion
Change of inflammation marker (hsCRP) | 3 months after electrical cardioversion
  Other markers can be added
Number of Participants with Adverse Events (AEs) | Participants will be followed for the duration of this study, an expected average 14 weeks
  All participants and practitioners are taught to report any AEs. If there are any AEs, the following items are recorded by practitioners at each visit and appropriate actions are taken: type of AEs, occurrence date, lost date, frequency of occurrence, severity, causality with the treatment, actions taken with the acupuncture intervention, and actions taken to the participants. Serious AEs, i.e. death or life-threatening events which are required urgent intervention, will be noted to the principal investigators immediately and determine whether the participants are dropped out.
the factor to make atrial fibrillation recur | 3 months later after electrical cardioversion
  we will perform multivariate regression analysis to know which factor makes atrial fibrillation recur irrespective of intervention method.

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, Professor, Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Kyung Hee University Medical Center, Seoul, Dongdaemun-gu, South Korea

REFERENCES:
- [Derived] Lee SM, Leem J, Park JH, Yoon KH, Woo JS, Lee JM, Kim JB, Kim W, Lee S. Close look at the experiences of patients enrolled in a clinical trial of acupuncture treatment for atrial fibrillation in Korea: a qualitative study nested within a randomised controlled trial. BMJ Open. 2017 Feb 3;7(2):e013180. doi: 10.1136/bmjopen-2016-013180. PMID 28159849
- [Derived] Park J, Kim HS, Lee SM, Yoon K, Kim WS, Woo JS, Lee S, Kim JB, Kim W. Acupuncture antiarrhythmic effects on drug refractory persistent atrial fibrillation: study protocol for a randomized, controlled trial. Evid Based Complement Alternat Med. 2015;2015:613970. doi: 10.1155/2015/613970. Epub 2015 Feb 17. PMID 25784948